CLINICAL TRIAL: NCT07182903
Title: Fatigue in MS: From Invisible to Measurable
Acronym: FIMS
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: UHasselt (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19721
Record Dates: First submitted 2025-09-03; First posted 2025-09-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; fatigue; cytotoxic CD4 T cells
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS: Participants with multiple sclerosis

SUMMARY:
Fatigue is one of the most common and burdensome symptoms of MS, but its precise cause remains unknown, and an effective treatment is lacking. Previous research has shown that the progression of MS is associated with a higher presence of a specific type of T-cell, the cytotoxic CD4+ T-cells, which play a role in the immune system.

The aim of this study is to investigate whether these cells can also be linked to fatigue in people with MS.

DETAILED DESCRIPTION:
Forty individuals with MS will be asked to complete questionnaires about fatigue and perform motor tasks. Additionally, blood samples will be taken to measure the levels of cytotoxic CD4+ T-cells. These values will then be correlated with fatigue scores and performance on the motor tasks.

Scores from the fatigue questionnaires and decline in amplitude and frequency from the performance fatiguability test will be correlated to the level of CD4 CTLs from the blood samples. Secondary study parameters include muscle activation patterns measured by EMG, distance walked on 6MWT and voluntary muscle activation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remittion, primary progressive or secondary progressive MS
* Age: 18-60 years
* Ability to perform the foot-tapping task
* Ability to walk at least 20 meters (with or without walking aid)

Exclusion Criteria:

* Dimethyl fumarate, fingolimod or alemtuzumab treatment, since these medications have a strong influence on the immune system As a result of these treatments, there are few to no immune cells circulating in the blood, meaning we cannot find our population of interest in the blood.
* Change in medication 6 weeks before the start of the study (including medication not related to MS) - MS relapse within 6 weeks of the start of the study
* Had an infection in the last month - Received a vaccination in the last 14 days - Pregnant or pregnancy in the last 6 months
* Having a psychiatric disorder
* Having a neurological disorder other than MS
* Having cognitive or communicative problems that makes it hard to follow instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 40 pwMS
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between percentage of cytotoxic CD4+ T cells and FSS score | Day 1
  Bivariate correlations will be calculated between the percentage of cytotoxic CD4+ T cells and fatigue, measured with Fatigue Severity Scale (FSS).
Correlation between percentage of cytotoxic CD4+ T cells and MFIS score | Day 1
  Bivariate correlations will be calculated between the percentage of cytotoxic CD4+ T cells and fatigue, measured with Modified Fatigue Impact Scale (MFIS).
Correlation between percentage of cytotoxic CD4+ T cells and foot-tapping frequency decrease | Day 1
  Bivariate correlations will be calculated between the percentage of cytotoxic CD4+ T cells and fatigability, measured as the decrease in frequency from the first 10 seconds of the task to the last 10 seconds of the task.
Correlation between percentage of cytotoxic CD4+ T cells and foot-tapping amplitude decrease | Day 1
  Bivariate correlations will be calculated between the percentage of cytotoxic CD4+ T cells and fatigability, measured as the decrease in amplitude from the first 10 seconds of the task to the last 10 seconds of the task.

SECONDARY OUTCOMES:
Changes in muscle activation during 6MWT | Day 1
  Comparison of the root-mean-square (RMS) of the EMG signal at the beginning of the task and the end of the task.
Changes in muscle activation during foot tapping task | Day 1
  Comparison of the root-mean-square (RMS) of the EMG signal at the beginning (first 10 seconds) of the task and the end (last 10 seconds) of the task.
Correlation changes in walking distance between the first and last minute of the 6MWT and CD4+ CTLs | Day 1
  Changes in distance between the first minute and the last minute of the 6MWT are measured to assess walking fatigability and will be correlated with the percentage of CD4+ CTLs in the blood.
Correlation percentage voluntary muscle activation and CD4+ CTLs | Day 1
  The correlation is calculated between the percentage of CD4+ CTLs in the blood and the percentage of voluntary activation (1 - superimposed twitch/initial-doublet) x 100%).

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided